CLINICAL TRIAL: NCT04434274
Title: Efficacy of MIcronized Purified Flavonoid Fraction-Based Phlebotropic Therapy After Endovenous MechanO-Chemical Ablation
Brief Title: MIcronized Flavonoid Fraction After MechanO-Chemical Ablation
Acronym: MIFFMOCA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Belarusian State Medical University (Other)
Responsible Party: Principal Investigator, Vladimir Khryshchanovich, Professor, Belarusian State Medical University
Other Study IDs: 20140455
Record Dates: First submitted 2020-06-10; First posted 2020-06-16 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Varicose Veins; Surgery
Keywords: VV; MPPF; MOCA; QoL
MeSH Terms: conditions — Varicose Veins

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A, MPFF-group: MPFF [Detralex®, Servier, France] 1,000 mg OD for 30 days in the postoperative period.
  Interventions: Drug: Micronized Purified Flavonoid Fraction
- Group B: No venoactive drug prescribed in the postoperative period.

INTERVENTIONS:
Drug: Micronized Purified Flavonoid Fraction — Based on the (non-)use of adjuvant phlebotropic therapy in the postoperative period.
  Other Names: Endovenous Mechano-Chemical Ablation
  Groups: Group A, MPFF-group

SUMMARY:
This study will be evaluate the clinical efficacy of micronized purified flavonoid fraction (MPFF) phlebotropic therapy for postoperative pain, venospecific symptoms, and quality of life in patients with incompetent great or small saphenous veins (GSV/SSV) following an endovenous mechanochemical ablation procedure (MOCA).

DETAILED DESCRIPTION:
The pre-op examination involved taking patient history (including the information about prior venous surgeries), identifying varicose veins (VV's) clinical symptoms/signs, duplex ultrasound (US) evaluation of the lower extremities, clinical-etiological and anatomical-pathophysiological assessment based on the CEAP classification.

The primary transverse and longitudinal US examination (B-mode, color and spectral Doppler) was performed by expert doctors at the Vascular Pathology Non-Invasive Diagnostics Unit before deciding on treatment choices. Reflux in the saphenofemoral/saphenopopliteal junction (SFJ/SPJ) area was determined in supine and upright positions using the Valsalva manoeuvre or manual compression/decompression test, respectively. SFJ/SPJ and great/small saphenous vein (GSV/SSV) segments with retrograde blood flow longer than 0.5 seconds were considered incompetent. Venous reflux section length and incompetent GSV/SSV segments' diameter (in mm) were reflected in medical documentation.

The trial inclusion criteria were as follows: age >18 years old; VV's CEAP clinical class C2-C4; SFJ/SPJ insufficiency and pathological (>0.5 s) reflux in GSV/SSV manifested by one or more "venous" symptoms (pain, itching, nocturnal leg cramps, swelling/pulsing sensation, heaviness, fatigue and overall discomfort), vein diameter at the SFJ/SPJ >4.5 mm and <8 mm in an upright position.

The patients were informed about the MOCA technique, the intervention's potential complications and side effects.

The exclusion criteria included isolated reflux in tributaries, excessive GSV/SSV tortuosity, known allergy to the sclerosant, deep/superficial vein thrombosis, post-thrombotic occlusion, confirmed thrombophilia, postoperative VV recurrence, obliterating peripheral artery diseases (ankle-brachial pressure index <0.8), pregnancy and lactation.

The Flebogrif™ device's design is based on a 5Fr single-channel diagnostic vascular catheter 60 cm or 90 cm long (with 1-cm graduated marks), its lumen containing a retractable metal rod with five sharp wires ("claws") attached to its tip. As the "claws" get released and the catheter is then withdrawn from the vessel, the vein wall's endothelial layer gets damaged; at this time, the distance between the fully opened cutting elements is ~29 mm, which is quite enough to treat incompetent veins up to 17-20 mm in diameter.

The patients were put in supine or prone positions for GSV or SSV ablation, respectively. The catheter length choice was determined by that of the incompetent vein segment. The GSV/SSV was punctured with a straight needle 18G at the distal point of reflux in an operating room under local anesthesia (1% lidocaine hydrochloride solution) and US guidance, after which a 0.035" J-shape guidewire was employed to insert a 6Fr introducer with an expander. Upon the latter's removal, a Flebogrif™ catheter was delivered to the target vein's lumen so as to have its tip positioned 2-3 cm below the SFJ/SPJ. Following the guidewire's removal, the catheter's cutting elements were released, shifting its outer "shell" against the stationary inner rod, after which a syringe containing a dose of 3% lauromacrogol-400 foamed solution (Ethoxysclerol®, Kreussler & Co. GmbH, Wiesbaden, Germany) prepared using the Tessari's method was connected to the central channel's port. The catheter was being distally removed from the vein in a smooth motion all the way up to the introducer, damaging the endothelium with its cutters, with simultaneous introduction of the foam in the amount of 0.1-0.2 ml per 1 cm. The graduated marks on the catheter helped measure the treated GSV/SSV section's length. During and within 5 minutes after the foam injection, the ultrasound probe was used to apply percutaneous compression in the SFJ/SPJ plane. Where deemed necessary, MOCA was supplemented with simultaneous Müller- Varadi miniphlebectomy or standard foam sclerotherapy of the visible varicose tributaries.

Immediately after the procedure, a class 2 RAL compression stocking was put on the operated lower limb, and the patients were recommended a 30-minute walk. The duration of elastic compression was continuous over the first 24 hours, with subsequent transition to daytime wear for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Great and small saphenous vein (GSV/SSV) incompetence with reflux at least down to the knee level.
2. Primary symptomatic varicose veins, Clinical Etiological Anatomical Pathophysiological (CEAP) classification, clinical class C2-C4.
3. Physical status according to American Society of Anesthesiologists (ASA) I-II (I-Healthy, non-smoking, no or minimal alcohol use; II-Mild diseases only without substantive functional limitations).
4. Ability to comprehend and sign an informed consent document.

Exclusion Criteria:

1. Postoperative varicose veins disease recurrence.
2. Deep venous thrombosis, thrombophilia associated with a high risk of deep venous thrombosis or postthrombotic syndrome.
3. Arterial occlusive disease more severe than Intermittent claudication after more than 200 meters of pain free walking (Fontaine IIA) and/or ankle brachial index below 0.8.
4. History of pulmonary embolism or stroke.
5. Current anticoagulation therapy (within 7 days of enrollment).
6. Pregnant or lactating women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with GSV/SSV incompetence and C2-C4 were included in in the prospective consecutive case study if they satisfied the selection criteria
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-06-18 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with pain from absent (score 0) to severe (score 3) | 7 days
  None (0), Occasional (1), Daily, interfering with, but not preventing regular daily activities (2), Daily, limiting most regular daily activities (3)
Number of Participants with pain from absent (score 0) to severe (score 3) | 14 days
  None (0), Occasional (1), Daily, interfering with, but not preventing regular daily activities (2), Daily, limiting most regular daily activities (3)
Number of Participants with pain from absent (score 0) to severe (score 3) | 30 days
  None (0), Occasional (1), Daily, interfering with, but not preventing regular daily activities (2), Daily, limiting most regular daily activities (3)
Number of Participants with other discomfort (ie aching, heaviness, fatigue, soreness, burning) from absent (score 0) to severe (score 3) | 7 days
  None (0), Occasional (1), Daily, interfering with, but not preventing regular daily activities (2), Daily, limiting most regular daily activities (3)
Number of Participants with other discomfort (ie aching, heaviness, fatigue, soreness, burning) from absent (score 0) to severe (score 3) | 14 days
  None (0), Occasional (1), Daily, interfering with, but not preventing regular daily activities (2), Daily, limiting most regular daily activities (3)
Number of Participants with other discomfort (ie aching, heaviness, fatigue, soreness, burning) from absent (score 0) to severe (score 3) | 30 days
  None (0), Occasional (1), Daily, interfering with, but not preventing regular daily activities (2), Daily, limiting most regular daily activities (3)
Number of Participants with venous oedema from absent (score 0) to severe (score 3) | 7 days
  None (0), Limited to foot or ankle (1), Extends above ankle but below knee (2), Extends to knee or above (3)
Number of Participants with venous oedema from absent (score 0) to severe (score 3) | 14 days
  None (0), Limited to foot or ankle (1), Extends above ankle but below knee (2), Extends to knee or above (3)
Number of Participants with venous oedema from absent (score 0) to severe (score 3) | 30 days
  None (0), Limited to foot or ankle (1), Extends above ankle but below knee (2), Extends to knee or above (3)
Number of Participants with inflammation from absent (score 0) to severe (score 3) | 7 days
  None (0), Limited to paramalleolar area (1), Diffuse over lower third of calf (2), Wider distribution (above lower third of calf) (3)
Number of Participants with inflammation from absent (score 0) to severe (score 3) | 14 days
  None (0), Limited to paramalleolar area (1), Diffuse over lower third of calf (2), Wider distribution (above lower third of calf) (3)
Number of Participants with inflammation from absent (score 0) to severe (score 3) | 30 days
  None (0), Limited to paramalleolar area (1), Diffuse over lower third of calf (2), Wider distribution (above lower third of calf) (3)

SECONDARY OUTCOMES:
Responders to Treatment, Assessed by Duplex Ultrasound | 8 weeks
  Responders; elimination of reflux through the saphenofemoral/saphenopopliteal junctions and/or coplete occlusion of the great/small saphenous veins at 8 weeks, as measured by duplex ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Khryshchanovich, MD, Prof, Study Chair — Educational Institution "Belarusian State Medical University"
Locations (1):
- Educational Institution "Belarusian State Medical University", Minsk, Dzerzhinski Ave., 83,, Belarus

IPD SHARING:
Plan to Share IPD: Yes
To evaluate clinical efficacy of micronized purified flavonoid fraction (MPFF) phlebotropic therapy for postoperative pain, venospecific symptoms, and quality of life in patients with varicose veins (VV) following an endovenous mechanochemical ablation procedure (MOCA).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 12.2020
Access Criteria: To evaluate clinical efficacy of micronized purified flavonoid fraction (MPFF) phlebotropic therapy for postoperative pain, venospecific symptoms, and quality of life in patients with varicose veins (VV) following an endovenous mechanochemical ablation procedure (MOCA).

REFERENCES:
- [Background] Nicolaides AN. The Benefits of Micronized Purified Flavonoid Fraction (MPFF) Throughout the Progression of Chronic Venous Disease. Adv Ther. 2020 Feb;37(Suppl 1):1-5. doi: 10.1007/s12325-019-01218-8. Epub 2020 Jan 22. PMID 31970659
- [Background] Pokrovsky AV, Saveljev VS, Kirienko AI, Bogachev VY, Zolotukhin IA, Sapelkin SV, Shvalb PG, Zhukov BN, Vozlubleny SI, Sabelnikov VV, Voskanian YE, Katelnitsky II, Burleva EP, Tolstikhin VY. Surgical correction of varicose vein disease under micronized diosmin protection (results of the Russian multicenter controlled trial DEFANS). Angiol Sosud Khir. 2007;13(2):47-55. English, Russian. PMID 18004259
- [Background] Bogachev VIu, Golovanova OV, Kuzhetsov AN, Shekoian AO. [On advisability of perioperative phleboprotection in endovascular treatment of lower in varicose disease: first initial results of the decision study]. Angiol Sosud Khir. 2012;18(2):90-5. Russian. PMID 22929677
- [Background] Bogachev VY, Boldin BV, Lobanov VN. Benefits of micronized purified flavonoid fraction as adjuvant therapy on inflammatory response after sclerotherapy. Int Angiol. 2018 Feb;37(1):71-78. doi: 10.23736/S0392-9590.17.03868-8. Epub 2017 Sep 22. PMID 28945060
- [Background] Mansilha A, Sousa J. Benefits of venoactive drug therapy in surgical or endovenous treatment for varicose veins: a systematic review. Int Angiol. 2019 Aug;38(4):291-298. doi: 10.23736/S0392-9590.19.04216-0. Epub 2019 Jul 5. PMID 31284708
- [Background] Sun JJ, Chowdhury MM, Sadat U, Hayes PD, Tang TY. Mechanochemical Ablation for Treatment of Truncal Venous Insufficiency: A Review of the Current Literature. J Vasc Interv Radiol. 2017 Oct;28(10):1422-1431. doi: 10.1016/j.jvir.2017.07.002. Epub 2017 Aug 12. PMID 28811080